CLINICAL TRIAL: NCT04131166
Title: Precision Nutrition and Metabolic Function
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Centene Corporation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 201908237
Record Dates: First submitted 2019-10-15; First posted 2019-10-18 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Obesity; Insulin Resistance
MeSH Terms: conditions — Obesity; Insulin Resistance | interventions — Diet, Mediterranean; Diet, Ketogenic; Diet, Fat-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Metabolically healthy lean (Other): Metabolically normal lean - Lean individuals that have good glucose (sugar) control, normal plasma triglyceride (fat) levels and a low liver fat content.
  Interventions: Other: Annual follow-up testing for 5 years
- Metabolically healthy obese - Mediterranean diet (Experimental): Metabolically normal obese - Persons with obesity that have good glucose (sugar) control, normal plasma triglyceride (fat) levels and a low liver fat content randomized to the Mediterranean diet group.
  Interventions: Behavioral: Mediterranean diet; Other: Annual follow-up testing for 5 years
- Metabolically healthy obese - Low-carbohydrate ketogenic diet (Experimental): Metabolically normal obese - Persons with obesity that have good glucose (sugar) control, normal plasma triglyceride (fat) levels and a low liver fat content randomized to the low-carbohydrate ketogenic diet group.
  Interventions: Behavioral: Low-carbohydrate, ketogenic diet; Other: Annual follow-up testing for 5 years
- Metabolically normal obese - Low-fat diet (Experimental): Metabolically normal obese - Persons with obesity that have good glucose (sugar) control, normal plasma triglyceride (fat) levels and a low liver fat content randomized to the low-fat diet group.
  Interventions: Behavioral: Low-fat diet; Other: Annual follow-up testing for 5 years
- Metabolically unhealthy obese - Mediterranean diet (Experimental): Metabolically abnormal obese - Persons with obesity with glucose levels higher than recommended and a moderate to high amount of fat in the liver randomized to the Mediterranean diet group.
  Interventions: Behavioral: Mediterranean diet; Other: Annual follow-up testing for 5 years
- Metabolically unhealthy obese - Low-carbohydrate ketogenic diet (Experimental): Metabolically abnormal obese - Persons with obesity with glucose levels higher than recommended and a moderate to high amount of fat in the liver randomized to the low-carbohydrate, ketogenic diet group.
  Interventions: Behavioral: Low-carbohydrate, ketogenic diet; Other: Annual follow-up testing for 5 years
- Metabolically unhealthy obese - Low-fat diet (Experimental): Metabolically abnormal obese - Persons with obesity with glucose levels higher than recommended and a moderate to high amount of fat in the liver randomized to the low-fat diet group.
  Interventions: Behavioral: Low-fat diet; Other: Annual follow-up testing for 5 years

INTERVENTIONS:
Behavioral: Mediterranean diet — A Mediterranean-type diet will be consumed for 4 to 8 weeks in the weight stable state with all meals provided.
  Arms: Metabolically healthy obese - Mediterranean diet; Metabolically unhealthy obese - Mediterranean diet
Behavioral: Low-carbohydrate, ketogenic diet — A low-carbohydrate, ketogenic diet will be consumed for 4 to 8 weeks in the weight stable state with all meals provided.
  Arms: Metabolically healthy obese - Low-carbohydrate ketogenic diet; Metabolically unhealthy obese - Low-carbohydrate ketogenic diet
Behavioral: Low-fat diet — A low-fat diet will be consumed for 4 to 8 weeks in the weight stable state with all meals provided.
  Arms: Metabolically normal obese - Low-fat diet; Metabolically unhealthy obese - Low-fat diet
Other: Annual follow-up testing for 5 years — Annual follow-up testing with no restrictions on dietary intake during periods between annual testing.

SUMMARY:
The purposes of this study are: 1) to determine the mechanisms responsible for the development of cardiometabolic complications in some, but not all people with obesity; 2) determine the best dietary approach for cardiometabolic health; and 3) understand why some people have a stable metabolic phenotype over time whereas cardiometabolic health improves or worsens in others.

DETAILED DESCRIPTION:
Excess adiposity causes alterations in metabolic function including impaired glucose homeostasis and insulin resistance, which are important risk factors for type 2 diabetes (T2D) and cardiovascular disease (CVD). Not all people with obesity experience the typical metabolic complications associated with obesity. Approximately 25% of people with obesity are protected from the adverse metabolic effects of excess fat accumulation and are considered to be metabolically healthy based on their normal response to insulin. The mechanism(s) responsible for the differences in metabolic function among people with obesity is not known, but is likely to be multifactorial including dietary intake. The risk for developing T2D and CVD is also well known to increase with age, however, not all people that are metabolically healthy convert to a metabolically unhealthy phenotype over time. The mechanisms responsible for the stability of health status in some, but not all adults, are unclear. The overall goals of this study are to: i) determine the mechanisms responsible for the development of cardiometabolic complications in participants who will be carefully characterized into 3 distinct groups [metabolically normal lean, metabolically normal obese and metabolically abnormal obese], ii) to determine the optimal dietary approach for cardiometabolic health independent of weight change in people with metabolically abnormal obesity, and iii) perform a comprehensive longitudinal assessment of cardiometabolic health to understand why some people have a stable metabolic phenotype over time whereas cardiometabolic health improves or worsens in others.

ELIGIBILITY:
Inclusion Criteria:

* Metabolically healthy lean subjects must have a body mass index (BMI) 18.5-24.9 kg/m2, intrahepatic triglyceride (IHTG) content ≤5%, serum triglyceride (TG) concentration <150 mg/dl, fasting plasma glucose concentration <100 mg/dl, 2-hr oral glucose tolerance test (OGTT) plasma glucose concentration ≤140 mg/dl, and hemoglobin A1C (HbA1C) ≤5.6%.
* Metabolically healthy obese subjects must have a BMI 30-49.9 kg/m2; IHTG content ≤5%, serum TG concentration <150 mg/dl, fasting plasma glucose concentration <100 mg/dl, 2-hr OGTT plasma glucose concentration ≤140 mg/dl, and HbA1C ≤5.6%.
* Metabolically unhealthy obese subjects must have a BMI 30-49.9 kg/m2; IHTG content ≥5.6% and fasting plasma glucose concentration ≥100 mg/dl or 2-hr OGTT plasma glucose concentration ≥140 mg/dl or HbA1C ≥5.7%.

Exclusion Criteria:

* medical, surgical, or biological menopause;
* previous bariatric surgery where the gastrointestinal tract is reconstructed such as Roux-en-Y, sleeve gastrectomy and biliopancreatic diversion surgeries;
* laparoscopic adjustable gastric band (lab band) surgery within the last 3 years;
* structured exercise ≥250 min per week (e.g., brisk walking);
* unstable weight (>4% change during the last 2 months before entering the study);
* significant organ system dysfunction (e.g., diabetes requiring medications, severe pulmonary, kidney or cardiovascular disease);
* cancer or cancer that has been in remission for <5 years;
* polycystic ovary syndrome;
* major psychiatric illness;
* conditions that render subject unable to complete all testing procedures (e.g., severe ambulatory impairments, limb amputations, or metal implants that interfere with imaging procedures; coagulation disorders);
* severe anemia;
* regular use of tobacco products;
* excessive consumption of alcohol (≥3 drinks/day for men and ≥2 drinks/day for women);
* use of medications that are known to affect the study outcome measures (e.g., steroids, non-statin lipid-lowering medications) or increase the risk of study procedures (e.g., anticoagulants) and that cannot be temporarily discontinued for this study;
* use of antibiotics in last 60 days;
* pregnant or lactating women;
* vegans, vegetarians, those with lactose intolerance and/or severe aversions/sensitivities to eggs, fish, nuts, wheat and soy, and/or any individuals with food allergies that induce an anaphylactic response;
* persons who are not able to grant voluntary informed consent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-10-08 (Actual); Primary Completion 2029-10-01 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Insulin sensitivity | Baseline only (cross-sectional comparison of metabolically healthy lean, metabolically healthy obese and metabolically unhealthy obese subjects).
  Whole-body insulin sensitivity will be assessed by using the hyperinsulinemic-euglycemic clamp procedure
Change in insulin sensitivity | Before and after 4-8 weeks of weight maintenance in metabolically healthy and unhealthy obese subjects randomized to follow a Mediterranean, low-carbohydrate or low-fat diet
  Whole-body insulin sensitivity will be assessed by using the hyperinsulinemic-euglycemic clamp procedure
Change in insulin sensitivity | Performed annually for 5 years
  Whole-body insulin sensitivity will be assessed by using the hyperinsulinemic-euglycemic clamp procedure

SECONDARY OUTCOMES:
24-hour glucose concentrations | Baseline only (cross-sectional comparison of metabolically healthy lean, metabolically healthy obese and metabolically unhealthy obese subjects).
  Plasma glucose concentrations will be evaluated from frequent blood samples over a 24 h period
Change in 24-hour glucose concentrations | Before and after 4-8 weeks of weight maintenance in metabolically healthy and unhealthy obese subjects randomized to follow a Mediterranean, low-carbohydrate or low-fat diet
  Plasma glucose concentrations will be evaluated from frequent blood sampling over a 24 h period
Change in 24-hour glucose concentrations | Performed annually for 5 years
  Plasma glucose concentrations will be evaluated from frequent blood sampling over a 24 h period
24-hour hormone concentrations | Baseline only (cross-sectional comparison of metabolically healthy lean, metabolically healthy obese and metabolically unhealthy obese subjects).
  Plasma hormone concentrations will be evaluated from frequent blood sampling over a 24 h period
Change in 24-hour hormone concentrations | Before and after 4-8 weeks of weight maintenance in metabolically healthy and unhealthy obese subjects randomized to follow a Mediterranean, low-carbohydrate or low-fat diet
  Plasma hormone concentrations will be evaluated from frequent blood samples over a 24 h period
Change in 24-hour hormone concentrations | Performed annually for 5 years
  Plasma hormone concentrations will be evaluated from frequent blood samples over a 24 h period
β-cell function | Baseline only (cross-sectional comparison of metabolically healthy lean, metabolically healthy obese and metabolically unhealthy obese subjects).
  β-cell function will be assessed from a modified oral glucose tolerance test
Change in β-cell function | Performed annually for 5 years
  β-cell function will be assessed from a modified oral glucose tolerance test
Insulin clearance | Baseline only (cross-sectional comparison of metabolically healthy lean, metabolically healthy obese and metabolically unhealthy obese subjects).
  Insulin clearance will be assessed from a modified oral glucose tolerance test and hyperinsulinemic-euglycemic clamp procedure
Change in Insulin clearance | Performed annually for 5 years
  Insulin clearance will be assessed from a modified oral glucose tolerance test and hyperinsulinemic-euglycemic clamp procedure
Fat mass and fat free mass | Baseline only (cross-sectional comparison of metabolically healthy lean, metabolically healthy obese and metabolically unhealthy obese subjects).
  Fat mass and fat free mass will be assessed using dual-energy x-ray absorptiometry (DXA)
Change in fat mass and fat free mass | Before and after 4-8 weeks of weight maintenance in metabolically healthy and unhealthy obese subjects randomized to follow a Mediterranean, low-carbohydrate or low-fat diet
  Fat mass and fat free mass will be assessed using dual-energy x-ray absorptiometry (DXA)
Change in fat mass and fat free mass | Performed annually for 5 years
  Fat mass and fat free mass will be assessed using dual-energy x-ray absorptiometry (DXA)
Exosome-mediated intercellular signaling | Baseline only (cross-sectional comparison of metabolically healthy lean, metabolically healthy obese and metabolically unhealthy obese subjects).
  Signaling between cells and organs will be examined by isolating exosomes (small extracellular vesicles) from blood and adipose tissue
Change in exosome-mediated intercellular signaling | Before and after 4-8 weeks of weight maintenance in metabolically healthy and unhealthy obese subjects randomized to follow a Mediterranean, low-carbohydrate or low-fat diet
  Signaling between cells and organs will be examined by isolating exosomes (small extracellular vesicles) from blood and adipose tissue
Change in exosome-mediated intercellular signaling | Performed annually for 5 years
  Signaling between cells and organs will be examined by isolating exosomes (small extracellular vesicles) from blood and adipose tissue
Intrahepatic triglyceride content | Baseline only (cross-sectional comparison of metabolically healthy lean, metabolically healthy obese and metabolically unhealthy obese subjects).
  Intrahepatic triglyceride content will be assessed by magnetic resonance imagining (MRI)
Change in intra-hepatic triglyceride content | Before and after 4-8 weeks of weight maintenance in metabolically healthy and unhealthy obese subjects randomized to follow a Mediterranean, low-carbohydrate or low-fat diet
  Intra-hepatic triglyceride content will be assessed by magnetic resonance imagining (MRI)
Change in intra-hepatic triglyceride content | Performed annually for 5 years
  Intra-hepatic triglyceride content will be assessed by magnetic resonance imagining (MRI)
Abdominal adipose tissue volumes | Baseline only (cross-sectional comparison of metabolically healthy lean, metabolically healthy obese and metabolically unhealthy obese subjects).
  Abdominal subcutaneous and intra-abdominal adipose tissue volumes will be assessed by magnetic resonance imagining (MRI)
Change in abdominal adipose tissue volumes | Before and after 4-8 weeks of weight maintenance in metabolically healthy and unhealthy obese subjects randomized to follow a Mediterranean, low-carbohydrate or low-fat diet
  Abdominal subcutaneous and intra-abdominal adipose tissue volumes will be assessed by magnetic resonance imagining (MRI)
Change in abdominal adipose tissue volumes | Performed annually for 5 years
  Abdominal subcutaneous and intra-abdominal adipose tissue volumes will be assessed by magnetic resonance imagining (MRI)
Leg adipose tissue volumes | Baseline only (cross-sectional comparison of metabolically healthy lean, metabolically healthy obese and metabolically unhealthy obese subjects).
  Thigh and calf adipose tissue volumes will be assessed by magnetic resonance imagining (MRI)
Change in leg adipose tissue volumes | Before and after 4-8 weeks of weight maintenance in metabolically healthy and unhealthy obese subjects randomized to follow a Mediterranean, low-carbohydrate or low-fat diet
  Thigh and calf adipose tissue volumes will be assessed by magnetic resonance imagining (MRI)
Change in leg adipose tissue volumes | Performed annually for 5 years
  Thigh and calf adipose tissue volumes will be assessed by magnetic resonance imagining (MRI)
Gut microbiome | Baseline only (cross-sectional comparison of metabolically healthy lean, metabolically healthy obese and metabolically unhealthy obese subjects).
  Gut microbiota, meta-transcriptome (bacterial RNA sequencing to determine what proteins can be made by the microbiota) and the meta-metabolome (metabolites made by the microbiota) will be assessed
Change in gut microbiome | Before and after 4-8 weeks of weight maintenance in metabolically healthy and unhealthy obese subjects randomized to follow a Mediterranean, low-carbohydrate or low-fat diet
  Gut microbiota, meta-transcriptome (bacterial RNA sequencing to determine what proteins can be made by the microbiota) and the meta-metabolome (metabolites made by the microbiota) will be assessed
Change in gut microbiome | Performed annually for 5 years
  Gut microbiota, meta-transcriptome (bacterial RNA sequencing to determine what proteins can be made by the microbiota) and the meta-metabolome (metabolites made by the microbiota) will be assessed
Carotid artery intima media thickness | Baseline only (cross-sectional comparison of metabolically healthy lean, metabolically healthy obese and metabolically unhealthy obese subjects).
  Carotid artery intima media thickness will be assessed by ultrasound imaging
Change in carotid artery intima media thickness | Performed annually for 5 years
  Carotid artery intima media thickness will be assessed by ultrasound imaging
Cardiac structure and function | Baseline only (cross-sectional comparison of metabolically healthy obese and metabolically unhealthy obese subjects).
  Ultrasound techniques will be used to assess cardiac structure and function
Change in cardiac structure and function | Performed annually for 5 years in metabolically healthy obese and metabolically unhealthy obese subjects.
  Ultrasound techniques will be used to assess cardiac structure and function
Endothelial function | Baseline only (cross-sectional comparison of metabolically healthy lean, metabolically healthy obese and metabolically unhealthy obese subjects).
  Endothelial function will be assessed using a non-invasive device (EndoPat 2000) in response to reactive hyperemia.
Change in endothelial function | Performed annually for 5 years
  Endothelial function will be assessed using a non-invasive device (EndoPat 2000) in response to reactive hyperemia.
Arterial stiffness | Baseline only (cross-sectional comparison of metabolically healthy lean, metabolically healthy obese and metabolically unhealthy obese subjects).
  Arterial stiffness will be assessed using a non-invasive device (SphygmoCor)
Change in arterial stiffness | Performed annually for 5 years
  Arterial stiffness will be assessed using a non-invasive device (SphygmoCor)
Transcriptome in blood, muscle and adipose tissue | Baseline only (cross-sectional comparison of metabolically healthy lean, metabolically healthy obese and metabolically unhealthy obese subjects).
  The transcriptome (all RNA that are responsible for making proteins from DNA templates) will be evaluated by using RNA sequencing techniques
Change in transcriptome in blood, muscle and adipose tissue | Performed annually for 5 years
  The transcriptome (all RNA that are responsible for making proteins from DNA templates) will be evaluated by using RNA sequencing techniques

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Klein, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Mittendorfer B, Patterson BW, Smith GI, Yoshino M, Klein S. beta Cell function and plasma insulin clearance in people with obesity and different glycemic status. J Clin Invest. 2022 Feb 1;132(3):e154068. doi: 10.1172/JCI154068. PMID 34905513